CLINICAL TRIAL: NCT02094872
Title: Stand Up to Cancer Consortium Genomics-Enabled Medicine for Melanoma (G.E.M.M.): Using Molecularly-Guided Therapy for Patients With BRAF Wild-Type (BRAFwt) Metastatic Melanoma
Brief Title: Molecularly Targeted Therapy in Treating Patients With BRAF Wild-type Melanoma That is Metastatic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1408014446; NCI-2014-00670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); WIRB Pro #20140190 (Other: Western Institutional Review Board (WIRB)); WO #1-822810-1 (Other: Western Institutional Review Board (WIRB)); Invest #161467 (Other: Western Institutional Review Board (WIRB)); Study #1144561 (Other: Western Institutional Review Board (WIRB)); 2013-184 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Recurrent Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Molecular Targeted Therapy; Coal Tar; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (molecularly targeted therapy) (Experimental): Patients undergo collection of tissue and blood samples for DNA and RNA analysis via sequencing. Based on the results of the DNA and RNA analysis, patients receive molecularly targeted therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: cytology specimen collection procedure; Drug: MEK 162 therapy or molecularly targeted therapy; Procedure: therapeutic procedure; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Other: cytology specimen collection procedure — Undergo collection of tissue and blood samples
  Other Names: cytologic sampling
Drug: MEK 162 therapy or molecularly targeted therapy — molecularly targeted therapy, MEK 162 therapy
Procedure: therapeutic procedure
  Other Names: Therapeutic Interventions; Therapeutic Method; Therapeutic Technique; Therapy; TX
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies how well molecularly targeted therapy works in treating patients with melanoma that has spread to other parts of the body. Patients must have received or do not qualify for prior immunotherapy. Targeted therapy is a type of treatment that uses drugs or other substances to identify and attack specific types of cancer cells with less harm to normal cells. Molecularly targeted therapy works by treating patients with substances that kill cancer cells by targeting key molecules involved in cancer cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the difference in best overall response rate (BORR) between patients treated with MEK162 following personalized molecularly guided assignment vs. a historical BORR of 7% in this patient population.

SECONDARY OBJECTIVES:

I. To evaluate the safety of performing individualized drug therapy (including novel agents and commercially-available agents) in the context of a personalized medicine clinical trial.

II. To define the difference in progression free survival (PFS) between patients treated with MEK162 following personalized molecularly guided assignment vs. a historical PFS rate of 2 months in this patient population.

III. To continually assess data in real time so as to iteratively refine and standardize a set of statistical and informatics methodologies for matching treatments to the patient's tumor, based on the molecular profile.

OUTLINE:

Patients undergo collection of tissue and blood samples for deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) analysis via sequencing. Based on the results of the DNA and RNA analysis, patients receive molecularly targeted therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient with metastatic or locally advanced and unresectable BRAF wild-type melanoma who have either progressed following previous treatment of immunotherapy, or are not eligible for immunotherapy; pts. are defined as "BRAF wild-type" if they test negative for V600 mutations based on a Clinical Laboratory Improvement Amendments (CLIA) certified assay
* Patients must have tumor accessible by interventional radiology or surgical intervention and suitable for biopsy (BX) with 5-6 passes of a 16 or 18 gauge needle for core BX (defined as at least 1 cm^3 tumor/50 mg accessible for BX), and must agree to undergo up to two surgical resections/biopsies to collect tumor for research purposes; the first of these biopsies will occur at the beginning of the study, prior to genetic analysis and Rx; the second BX will be performed at the time of DZ progression/end of study should funding be available
* Patients must have measurable DZ (per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 [v1.1] criteria), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or a subcutaneous or superficial lesion that can be measured with calipers by clinical exam; for lymph nodes, the short axis must be >= 15 mm
* Previous therapies: prior radiation therapies, immunotherapies, and investigational therapies are allowed as follows.

  * Radiation: prior radiation therapy (RT) is allowed with the following conditions:

    * Patients who have received minimal RT (=< 5% of their total marrow volume) must have completed it >= 2 weeks prior to the initiation of study Rx
    * Patients who have received RT that constituted > 5% but < 50% of their total marrow volume must have completed it >= 4 weeks prior to the initiation of study treatment
    * Patients who have received prior radiation to 50% or more of their total marrow volume will be excluded
    * Patients may be biopsied while undergoing RT as long as BX site is not in the radiation portal; however, they still have to wait the required amount of time from radiation to treatment even though the tumor board may have already occurred and a treatment plan assigned
  * Other therapies: prior investigational or targeted therapies and immunotherapies may be allowed following discussion with the PI (PI); if the PI deems the prior treatment acceptable, patients must not have received these therapies for 28 days or five half-lives of the drug (whichever is lesser) prior to the initiation of study treatment and must have full recovery from any acute effects of these therapies; prior therapy with mitogen-activated protein kinase (MEK) inhibitors will not be allowed
* Patients with chronic grade 2 toxicity may be eligible at the discretion of the PI if the condition has been stable, and not worsening, for at least 30 days; pts. with ongoing alopecia of any grade will be eligible
* Patient must have a life expectancy of >= 3 months, as estimated by the treating oncologist
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin >= 9 g/dL
* Leukocytes >= 3,000/microliter (mcL)
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets (PLT) >= 100,000/mcL
* Aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN); if liver metastases are present, =< 5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN; if liver metastases are present, =< 5 x ULN
* Bilirubin =< 1.5 x ULN
* Creatinine =< 1.5 x ULN OR calculated or measured creatinine clearance >= 50 mL/min/1.73 m^2 for pts. with creatinine above institutional normal
* If available, pt. must agree to provide archival tissue for research purposes (either archival paraffin tissue block or 10 unstained slides of a primary or metastatic melanoma lesion) prior to enrollment; samples should be shipped within 1 month after enrollment
* Patient agrees to having a blood sample (a minimum of 10 mL, with 20 mL preferred) drawn and analyzed to compare their normal genetic profile to that of their tumor sample
* Patient must be able to tolerate oral medication
* Women of child-bearing potential and men must agree to use 2 forms of adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and for four months following completion of study therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; women who become pregnant must immediately discontinue Rx with any study therapy; male pts. should avoid impregnating a female partner; male pts., even if surgically sterilized, (i.e. post-vasectomy) must agree to one of the following: practice effective barrier contraception during the entire study Rx period and through 4 months after the last dose of study drug, or completely abstain from sexual intercourse
* Patient must have the ability to understand and the willingness to sign a written informed consent document
* Patient must be willing and able to comply with the protocol for the duration of the study, including attending scheduled visits, examinations, the BX procedure, and having their tumor and blood molecularly characterized
* Patient understands they must meet all inclusion and exclusion criteria in the drug specific appendix for which they were assigned.

Exclusion Criteria:

* Patients with peripheral neuropathy >= grade 2 are not permitted unless discussed with the PI and only in unique circumstances (i.e. unilateral neuropathy due to trauma)
* Patient has DZ that tests positive for BRAF V600 mutations based on the results of a CLIA certified assay
* Patients with active infection at time of BX
* Patients with any evidence of severe or uncontrolled systemic DZ(s) including known cases of hepatitis B or C or human immunodeficiency virus (HIV); screening for chronic conditions is not required, although pts. known to have such conditions at screening should not be included
* Any patient requiring chronic maintenance of red blood cell, white blood cell or granulocyte counts through the use of blood transfusions or growth factor support (e.g. Neulasta®, Neupogen®)
* Patients with a prior history of seizures within the past year unrelated to brain metastases
* Patients with known active progressive brain metastases; pts. with prior treated brain metastases are allowed, providing that they were not accompanied by seizures within the past year and that a baseline brain MRI scan prior to study entry demonstrates no current evidence of active brain metastases; all pts. with prior treated brain metastases must be stable for > 1 months after treatment and off steroid treatment prior to study enrollment
* Patients receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (i.e. megestrol acetate, bisphosphonates); these medications must have been started >= month prior to enrollment on this study; pts. may be on low molecular weight heparin or direct factor Xa inhibitors
* Patients with any clinically significant medical condition which, in the opinion of the investigator, makes it undesirable for the pt. to participate in the study or which could jeopardize compliance with protocol requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness/social situations
* Patients with preexisting cardiac conditions, including uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure will not be eligible
* Patients with left ventricular ejection fraction (LVEF) < 45% will not be eligible
* Patients with either of the following within 6 months before the first dose of study treatment:

  * Stroke (including transient ischemic attack [TIA], or other ischemic event)
  * Myocardial infarction
* Patients with acute gastrointestinal bleeding within 1 month of study entry
* Patients who have, at screening, corrected QT interval using Fridericia's formula (QTcF) >= 450 msec for males and QTcF >= 470 for females
* Patients with a co-morbid condition(s) that, in the opinion of the investigator, prevents safe surgery/BX procedure
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption or ability to swallow oral medication
* Pregnant or nursing women; breastfeeding must be discontinued prior to Rx
* Patients who have received organ transplant
* Patients who have had major surgery within 14 days of study enrollment
* Patients diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, or an in situ malignancy. Patients with a low grade prostate cancer, not on hormonal therapy, for which the disease is confined to the prostate may be considered eligible by the overall Principal Investigator on a case by case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-05; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, D.O., Principal Investigator — Yale University
Locations (8):
- United States (8):
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Sammons Cancer Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Based on the initial 23 patients enrolled on this study who underwent molecular profiling and tumor board evaluation, 20 were assigned MEK162 by the tumor board. Patients not assigned MEK162 still received their assigned treatment, but were not considered evaluable for the primary endpoint.
Groups:
- Arm I (Molecularly Targeted Therapy): Patients undergo collection of tissue and blood samples for DNA and RNA analysis via sequencing. Based on the results of the DNA and RNA analysis, patients receive molecularly targeted therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  cytology specimen collection procedure: Undergo collection of tissue and blood samples
  MEK 162 therapy or molecularly targeted therapy: molecularly targeted therapy, MEK 162 therapy
  therapeutic procedure
  laboratory biomarker analysis: Correlative studies
  quality-of-life assessment: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Molecularly Targeted Therapy)
Started | 49
Received Biopsy | 37
Received Tumor-board Recommendation | 36 (1 individual withdrew consent after biopsy.)
Received Targeted Therapy | 20
Received Standard of Care | 9 (7 standard-of-care patients crossed-over and received targeted therapy.)
Patients Treated With MEK162 (Total patients treated with MEK162 for final primary endpoint (following study redesign)) | 20
Completed | 20
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | Arm I (Molecularly Targeted Therapy)
Number analyzed (Participants) | 49
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 1
  40-49 | 6
  50-59 | 10
  60-69 | 13
  70-79 | 15
  80-89 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0
  Asian or Pacific Islander | 0
  Black, not of Hispanic Origin | 2
  Hispanic | 6
  White, not of Hispanic Origin | 43
  Other/ | 4
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR)
Description: The best overall response rate (BORR) was assessed up to 1 year.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Molecularly Targeted Therapy)
Number analyzed (Participants) | 20
Participants
  Progressive Disease | 2
  Stable Disease | 17
  Partial Response | 1

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: A log rank test will be performed for the comparison between the two groups.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
Population: Given the lack of response in this study and the decision to terminate it early, no data for PFS data were collected or analyzed. In addition, with the study amendment removing the second arm, this analysis would not have been possible to conduct.
Arm/Group | Arm I (Molecularly Targeted Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm I (Molecularly Targeted Therapy)
All-Cause Mortality (participants affected / at risk) | 5/49
Serious Adverse Events (participants affected / at risk) | 48/49
Other Adverse Events (participants affected / at risk) | 32/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Molecularly Targeted Therapy) (N=49)
Anaphylactic reaction to taxol, hospitalized (Immune system disorders) | 1
Allergic reaction to Augmentin; Acute kidney Injury (patient never received drug) (Immune system disorders) | 1
Acneiform rash (Skin and subcutaneous tissue disorders) | 1
Elevated alkaline phosphatase (Skin and subcutaneous tissue disorders) | 1
Elevated aspartate aminotransferase (Skin and subcutaneous tissue disorders) | 3
Elevated alanine aminotransferase (Skin and subcutaneous tissue disorders) | 1
Transaminitis (Skin and subcutaneous tissue disorders) | 1
Creatine phosphokinase elevation (Skin and subcutaneous tissue disorders) | 2
Uric acid elevations (Skin and subcutaneous tissue disorders) | 1
Hospitalized for hypotension related to adrenal insufficiency (Vascular disorders) | 1
Hospitalized for hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hospitalized for pulmonary embolism (Vascular disorders) | 3
Hypotensive, AKI (patient never received drug) (Vascular disorders) | 1
Generalized Weakness (General disorders) | 1
Fatigue (General disorders) | 2
Weakness and fatigue (General disorders) | 1
Hospitalized for generalized weakness (General disorders) | 1
Generalized weakness requiring hospitalization; outcome death (General disorders) | 1
Hospitalized for pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalized for pneumonia, sepsis, outcome death (Respiratory, thoracic and mediastinal disorders) | 1
Hospitalized for Nausea and vomiting (Gastrointestinal disorders) | 1
Anemia due to gastric hemorrhage (Gastrointestinal disorders) | 1
Hospitalized for abdominal and back pain (Gastrointestinal disorders) | 1
Hepatic Failure (patient never received drug) (Hepatobiliary disorders) | 1
Radical resection of malignant soft tissue tumor (melanoma) on back (Surgical and medical procedures) | 1
Hospitalized for anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hospitalized for chronic intractable pain (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hospitalization for neurological symptoms: brain metastasis (Nervous system disorders) | 1
Dropped Head Syndrome (Musculoskeletal and connective tissue disorders) | 1
Ocular muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hospitalized for back pain (Musculoskeletal and connective tissue disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypochloridemia (Metabolism and nutrition disorders) | 1
Hospitalized for UTI (Infections and infestations) | 1
Enterocolitis infectious (Clostridium difficile) (Infections and infestations) | 1
Hospitalized for fever (Infections and infestations) | 1
Strep B sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Molecularly Targeted Therapy) (N=49)
Anemia (Blood and lymphatic system disorders) | 11
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Endocrine disorders - Other (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Blurred vision (Eye disorders) | 2
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 6
Glaucoma (Eye disorders) | 1
retinal detachment (Eye disorders) | 1
watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 19
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 12
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 22
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Chills (General disorders) | 6
Edema face (General disorders) | 2
Fatigue (General disorders) | 25
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 3
Gait disturbance (General disorders) | 2
General disorders and administration site conditions - Other, specify (General disorders) | 12
Pain (General disorders) | 1
Edema limbs (General disorders) | 15
Infusion related reaction (General disorders) | 1
Localized edema (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 2
Cardiac troponin I increased (Investigations) | 1
Cardiac troponin T increased (Investigations) | 1
CPK increased (Investigations) | 10
Creatinine increased (Investigations) | 6
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 4
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
Weight gain (Investigations) | 3
Weight loss (Investigations) | 3
Hemoglobin increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 12
Hypersomnia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Movements involuntary (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 7
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 7
Hematuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4
Urinary frequency (Renal and urinary disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythroderma (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 16
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Because of the lack of clinical response, it was decided that enrollment should discontinue. Twenty patients who received MEK162 were evaluated for the primary outcome; secondary outcome was not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02094872/Prot_SAP_000.pdf